CLINICAL TRIAL: NCT03246919
Title: Ideal Time of Oxytocin Infusion During Cesarean Section
Acronym: I-TOPICS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left Loyola and Sub-I graduated.
Sponsor: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 209632
Record Dates: First submitted 2017-08-04; First posted 2017-08-11 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2019-08

CONDITIONS: Blood Loss, Surgical; Postpartum Hemorrhage; Bleed Pregnancy; Pregnancy Related; Cesarean Section Complications
MeSH Terms: conditions — Blood Loss, Surgical; Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind: Obstetricians, Anesthesiologists and patients will be blinded. Only nurses will be aware of timing of oxytocin administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Group A) (Placebo Comparator): One bag of 500 ml 0.9% NaCl (normal saline) will be hung by Anesthesia when the fetal anterior shoulder delivers. After the placenta is delivered, then one bag of 500 ml 0.9% NaCl with 30 units of Oxytocin (Oxytocin solution) will be hung by Anesthesia. This amount of fluid is part of standard of care.
  Interventions: Drug: Placebo
- Intervention (Group B) (Active Comparator): One bag of 500 ml 0.9% NaCl with 30 units of Oxytocin (Oxytocin solution) will be hung by Anesthesia when the fetal anterior shoulder delivers. After the placenta is delivered, then one bag of 500 ml 0.9% NaCl (normal saline) will be hung by Anesthesia. This amount of fluid is part of standard of care.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin is administered after delivery of the fetal anterior shoulder, rather than being administered after delivery of the placenta
  Other Names: Pitocin
  Arms: Intervention (Group B)
Drug: Placebo — Placebo will be administered after delivery of the placenta
  Arms: Control (Group A)

SUMMARY:
This study will evaluate if the timing of oxytocin administration in cesarean deliveries will affect the amount of maternal blood loss. Half of participants will receive oxytocin after delivery of the fetal anterior shoulder and the other half will receive oxytocin after delivery of the placenta. We hypothesize that administering oxytocin after delivery of the shoulder, will result in less overall maternal blood loss.

DETAILED DESCRIPTION:
Oxytocin is a routinely administered medication for both vaginal and cesarean deliveries in the third stage of labor, as part of standard of care in the United States. This medication helps to reduce overall blood loss, by functioning as a uterotonic. Currently evidence is lacking to direct timing of oxytocin administration in cesarean deliveries.

This study will evaluate both estimated and quantitative blood loss for both groups of patients. It will also compare the change from pre-operative to post-operative hemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarean section at Loyola Hospital
* Women who read and speak the English and/or Spanish language
* Women age 18 or older

Exclusion Criteria:

* Women who deliver vaginally
* Gestation under 37 weeks and 0 days
* Women with coagulopathies
* Multiple gestation pregnancies
* Antepartum hemorrhage for example abruption
* Placental abnormalities for example previa, accreta

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Total blood loss | At the completion of the surgery when patient is transferred to recovery from the operating room
  Both the estimated blood loss and quantitative blood loss will be determined

SECONDARY OUTCOMES:
Incidence of postpartum hemorrhage | At the completion of the surgery when patient is transferred to recovery from the operating room
  The number of women who lose 1,000 milliliters or more blood from cesarean delivery
Need for transfusion | In the immediate 24 hours post surgery
  The number of women who require a blood transfusion due to surgical blood loss
Change in pre-operative to post-operative hemoglobin levels | Baseline and Post operative day number 1
  Hemoglobin levels

CONTACTS AND LOCATIONS:
Overall Officials: Thaddeus Waters, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson KW Jr, Allbert JR, Schemmer GK, Elliot M, Humphrey A, Taylor J. A randomized controlled trial comparing oxytocin administration before and after placental delivery in the prevention of postpartum hemorrhage. Am J Obstet Gynecol. 2001 Oct;185(4):873-7. doi: 10.1067/mob.2001.117363. PMID 11641669
- [Background] Soltani H, Hutchon DR, Poulose TA. Timing of prophylactic uterotonics for the third stage of labour after vaginal birth. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD006173. doi: 10.1002/14651858.CD006173.pub2. PMID 20687079
- [Background] Fidan U, Keskin U, Ulubay M, Efendi Karaca R, Burcin Firatligil F, Goksen Kocagoz G, Ergun A. The effect of the use of oxytocin on blood loss during different postpartum periods. J Perinat Med. 2015 Jul;43(4):461-5. doi: 10.1515/jpm-2014-0111. PMID 24897394
- [Background] Oguz Orhan E, Dilbaz B, Aksakal SE, Altinbas S, Erkaya S. Prospective randomized trial of oxytocin administration for active management of the third stage of labor. Int J Gynaecol Obstet. 2014 Nov;127(2):175-9. doi: 10.1016/j.ijgo.2014.05.022. Epub 2014 Jul 17. PMID 25108586
- [Background] Dahlke JD, Mendez-Figueroa H, Rouse DJ, Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery: an updated systematic review. Am J Obstet Gynecol. 2013 Oct;209(4):294-306. doi: 10.1016/j.ajog.2013.02.043. Epub 2013 Mar 1. PMID 23467047
- [Background] Khan FA, Khan M, Ali A, Chohan U. Estimation of blood loss during Caesarean section: an audit. J Pak Med Assoc. 2006 Dec;56(12):572-5. PMID 17312645
- [Background] Anderson JM, Etches D. Prevention and management of postpartum hemorrhage. Am Fam Physician. 2007 Mar 15;75(6):875-82. PMID 17390600
- [Background] WHO Recommendations for the Prevention and Treatment of Postpartum Haemorrhage. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK131942/ PMID 23586122
- [Background] National Collaborating Centre for Women's and Children's Health. Caesarean section NICE Clinical Guideline. Royal College of Obstetricians and Gynaecologists
- [Background] Silverman, F. & Bornstein, E. Pharmacologic management of the third stage of labor. UpToDate. 2015